CLINICAL TRIAL: NCT00496444
Title: Phase I Study of Low-Dose Hypomethylating Agent Azacitidine Combined With the Histone Deacetylase Inhibitor Valproic Acid in Patients With Advanced Cancers
Brief Title: Azacytidine and Valproic Acid in Patients With Advanced Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0735
Record Dates: First submitted 2007-07-02; First posted 2007-07-04 (Estimated); Last update posted 2012-08-01 (Estimated); Status verified 2012-07

CONDITIONS: Advanced Cancers
Keywords: Advanced Cancers; Azacytidine; 5-Azacitidine; 5-aza; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816; Valproic Acid; Depakene
MeSH Terms: interventions — Azacitidine; Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Azacitidine + Valproic Acid (Experimental)
  Interventions: Drug: Azacitidine; Drug: Valproic Acid

INTERVENTIONS:
Drug: Azacitidine — Starting Dose 20 mg/m^2 administered subcutaneously (under the skin), daily, for ten days (Days 1 -10) of every 4 Week Cycle.
  Other Names: 5-Azacitidine; 5-aza; Vidaza; 5-AZC; AZA-CR; Ladakamycin; NSC-102816
Drug: Valproic Acid — Starting Dose 10 mg/Kg once daily by mouth, every day of 4 Week Cycle.
  Other Names: Depakene

SUMMARY:
Primary Objective:

1. To evaluate side effects and maximum tolerated dose of azacitidine and valproic acid in patients with advanced cancer.

Secondary Objectives:

1. To perform a preliminary assessment of the histone acetylation and DNA methylation effects of this combination on peripheral blood mononuclear cells (PBMC).
2. To assess the clinical anti-tumor activity (objective response including complete and partial responses) of this combination in patients with advanced cancer, in a descriptive fashion.

DETAILED DESCRIPTION:
Azacitidine is a new chemotherapy drug that is designed to destroy cancer cells at high doses. At low doses, it is designed to destroy some cancer cells as well as cause changes that may make cancer cells less harmful. Valproic acid is a drug that is used in every day practice in the treatment of seizures, migraine headache, and mood disturbance in bipolar disorders.

Before you can start receiving the study drug, you will have what are called "screening tests." These tests will help the doctor decide if you are eligible to take part in the study. You will have a complete physical exam, including routine blood tests (about 4 teaspoons). You may have to get either a CT scan or a MRI to measure your disease if you have not had one within 1 month. Women who are able to have children must have a negative blood-pregnancy test.

If you are found to be eligible to take part in this study, you will receive the study drug in "cycles." Cycles will generally be 4 weeks long but may be longer, depending on any side effects you experience from the azacitidine. During each cycle, you will receive azacitidine under the skin once each day for the first 10 days (Day 1 to Day 10). You will then have an 18-day break during which you will not receive azacitidine injections for the rest of the cycle. Additionally, you will take valproic acid pills by mouth, every day, starting the first day of the first cycle (Day 1 to Day 28). You will take valproic acid every day while on study without interruption.

The dose of azacitidine that you receive will depend on when you enroll in this study. You will be part of a study group "cohort" (6 patients will be enrolled in each cohort). All members of a cohort receive the same dose of azacitidine when they begin receiving the study drug. Each new cohort will receive a higher dose than the cohort before. The dose of azacitidine that you receive may be adjusted depending on how well you tolerate it. The starting dose of valproic acid is fixed for all the patients, but this dose may be adjusted by your physician based on the results of your blood work.

You will have a physical exam and blood tests (about 1 tablespoon each) every two weeks of the first two study drug cycles. For further cycles, you will have a physical exam and blood test only once a month. Your disease will be measured by CT scan or MRI after every 2 treatment cycles.

You may continue to receive the study drug on this study until your disease gets worse or intolerable side effects occur. After your participation in this study is over, you will receive follow-up care, as is standard of care for your disease.

This is an investigational study. The FDA has approved azacitidine for a blood disease known as myelodysplastic syndrome. Its use in this study is experimental. The valproic acid is a drug approved by the FDA for treatment of seizure, bipolar disorders, and migraine headaches. Up to 68 patients will take part in the study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologically confirmed malignancy that is metastatic or unresectable and refractory to standard therapy or for whom there is no standard therapy that induces complete remission (CR) of at least 10% or an increased survival of at least 3 months.
2. There is no maximum allowable number of prior chemotherapy regimens, provided all other eligibility criteria are met.
3. No chemotherapy, radiotherapy, investigational agents or surgery within four weeks.
4. ECOG performance status 2 or less.
5. Normal organ and marrow function - ANC > 1500/microL - Platelets > 100,000/microL - Total bilirubin < 2.0 mg/dL - Creatinine < 2.0 mg/dL
6. The effect of azacytidine on the development of human fetus is unknown. Because of the chemotherapy agents are known to be teratogenic, women and men of childbearing potential must agree to use adequate contraception prior to study entry and for the duration of the study.
7. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Uncontrolled concurrent illness such as neutropenic fever,shock, symptomatic congestive heart failure (NYHA class III or IV).
2. Hypersensitivity to divalproex sodium, valproic acid, or valproate sodium
3. Known or suspected hypersensitivity to azacitidine or mannitol.
4. Nursing and pregnant women.
5. Patients with urea cycle disorders (UCD): - History of unexplained coma, encephalopathy, or mental retardation - Encephalopathy associated with a protein load - Pregnancy-related or postpartum encephalopathy - History of elevated plasma ammonia or glutamine - Those with cyclical vomiting and lethargy, episodic extreme irritability, ataxia, low BUN, or protein avoidance. - Those with a family history of UCD or unexplained infant deaths (particularly males).
6. Patients with a known ornithine transcarbamylase disorder, history of unexplained coma or a family history of ornithine transcarbamylase disorder are excluded from this study.
7. Patients younger than 2-year old since valproic acid safety is not proven in this age group.
8. Leukemias and MDS are excluded

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2005-05; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
To find the highest safe dose of the drug azacitidine that can be given in combination with valproic acid in the treatment of solid tumors. | 4 Years

CONTACTS AND LOCATIONS:
Overall Officials: Razelle Kurzrock, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- U.T.M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org